CLINICAL TRIAL: NCT01289197
Title: Health Promotion in Early Adolescence: Sleep, Activity, and Emotion Regulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Daniel Shaw, Principal Investigator, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 5R01HD057893-02 (NIH)
Record Dates: First submitted 2011-02-01; First posted 2011-02-03 (Estimated); Last update posted 2016-01-11 (Estimated); Status verified 2016-01

CONDITIONS: Sleep Disorders; Physical Activity; Depression; Anxiety
MeSH Terms: conditions — Sleep Wake Disorders; Motor Activity; Depression; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- No Feedback or services offered. (No Intervention): The Family Check-Up is not offered.
- Intervention (Other): Family Check Up is offered.
  Interventions: Behavioral: Family Check Up

INTERVENTIONS:
Behavioral: Family Check Up — Families in the intervention condition will be contacted by the parent consultant following the T1 and T2 assessments and be invited to participate in the Family Check-Up (FCU). The FCU intervention involves at least three sessions in which we expect both mother and child to participate in. First is the in-home family assessment. The second session involves rapport-building via an initial interview with the caregiver(s), referred to as the Get-to-Know-You visit, or for families already enrolled in an ongoing study, a Check-Back-In visit. The third is a Feedback Session during which the results of the assessment and initial interview are discussed with the caregiver, with attention focused on the caregiver's and child's readiness to change and the delineation of specific change options.
  Other Names: Sleeping Tigers; Project MOVE
  Arms: Intervention

SUMMARY:
The primary goal of this project is to examine the short and long-term effects of an intervention focusing on three interrelated dimensions of health: improving sleep, increasing physical activity, and improving skills in emotion regulation. This intervention targets high-risk youth at a key neuromaturational period-early adolescence-when many individuals are experiencing new challenges to regulatory systems involved in sleep, activity, and emotion regulation. This maturational period is also a crucial time in the normal development of habits, skills, and proclivities in each of these domains. Thus, early adolescence presents unique opportunities for intervention targeting these three interrelated regulatory systems. Participants will include 200 9-13 year-old children who are siblings of children enrolled in one of three ongoing studies of vulnerability and resilience, whose families were initially identified on the basis of sociodemographic, child, and/or family risk or are recruited thru local Family Centers. Children will be selected as having difficulties in at least one of these domains (sleep, sedentary behavior, or emotion regulation) and then randomly assigned to either a control or intervention group. All families will receive baseline, one- and two-year follow-up assessments of child sleep, physical activity, and emotion regulation. Families in the intervention group will have the opportunity to receive feedback and intervention services on these three child domains and other parenting and family issues (e.g., parent involvement, parent self-care, school problems) following the initial assessment and the one-year follow up. The intervention will involve the parent and target youth receiving feedback about the child's current status in these areas and family functioning. If desired, the family will also participate in follow-up meetings with the parent and/or target youth to improve the youth's sleep, physical activity, and/or emotion regulation skills, as well as aspects of the family environment. The investigators hypothesize that the intervention will be associated with improvements in sleep, physical activity, and emotion regulation among those in the intervention group, as well as improvements in measures of social, behavioral, and affective function. Finally, the investigators will explore the possibility that increases in parental involvement mediate some of the changes found in child sleep, physical activity, and emotion regulation.

DETAILED DESCRIPTION:
The primary objective of this project is to examine the short and long-term effects of an intervention focusing on three interrelated dimensions of health: improving sleep, increasing physical activity, and improving skills in emotion regulation. This intervention targets high-risk youth at a key neuromaturational period-early adolescence-when many individuals are experiencing new challenges to regulatory systems involved in sleep, activity, and emotion regulation.

SPECIFIC AIMS:

1. To examine the effects of the intervention on sleep, physical activity, and emotion regulation:

   Hypothesis 1a: The intervention will result in increased total sleep and more regularized sleep/wake schedules (as measured by Sensewear sleep/activity monitors and sleep logs in the home environment).

   Hypothesis 1b: The intervention will result in increased physical activity and less time per week in sedentary activity (as measured by Sensewear activity monitors and standardized physical activity questionnaire).

   Hypothesis 1c: The intervention will result in improved emotion regulation (as measured by a composite index derived from interaction tasks, as well as home and school measures of emotion regulation).
2. To examine intervention effects on externalizing (problem behavior), internalizing symptoms, and peer relationships.

   Hypothesis 2a: The intervention will result in lower levels of externalizing and internalizing symptoms and improved relationships with peers as measured by parent, youth, and teacher reports.

   Hypothesis 2b: Intervention effects for lower levels of externalizing and internalizing symptoms and improved relationships with peers, if found, will be mediated by improvements in child sleep, physical activity, and emotion regulation.

   SECONDARY AIMS: In addition to these specific aims the following exploratory analyses are planned:
3. To examine parent-child interaction as a mediator of change in child sleep, physical activity, and emotion regulation. Just as we are interested in the possibility that changes in child problem behavior and peer relationships are mediated by improvements in sleep, physical activity, and emotion regulation, we will examine aspects of improvements in sleep, physical activity, and emotion regulation that are mediated by improvements in the quality of parent-child interaction (e.g., parental involvement), based on both parent reports and observations of parent-child quality.
4. To explore directional effects between sleep, daytime activity, daytime mood, emotion regulation, and affective and behavioral symptoms. For example, we will examine: a) if sleep difficulties will predict daytime measures of negative mood, irritability, and decreased physical activity the following day; or b) if daytime measures of stress and negative affect will predict sleep difficulties the subsequent night; c) if physical activity during the day will be associated with better sleep that night.
5. To examine the impact of this intervention on measures of physical health (e.g., Body Mass Index and waist circumference) and academic function (e.g., days of school missed/tardiness and school performance).

ELIGIBILITY:
Inclusion Criteria:

* Eligibility in the study will be based on multiple criteria, including the family's low SES status (i.e., income less than 50% over the poverty line and no more than 2 years of college education for parents)
* Risk status on child problems with sleep, physical activity, and/or affect regulation. Criteria for the latter will be established using a 14-item screening procedure administered to parents.

Exclusion Criteria:

* Children or parents with severe mental health concerns that prohibit them from completing the assessment protocol or potentially benefiting from the intervention will not be eligible for participation (e.g., parents or children with severe mental retardation, autism, schizophrenia, or other psychotic disorders).
* If a child has a previous diagnosis of obstructive sleep apnea, they will still benefit from participating in the study and will not be excluded.
* Adolescents who are currently incarcerated or who are in a court mandated facility will be excluded from enrolling in the study.
* If an adolescent becomes incarcerated or is placed in a court mandated facility after enrollment in the study, he/she will be withdrawn from the study if the duration of incarceration or court mandated placement is longer than the amount of time remaining for study participation.
* However, adolescents who are transiently incarcerated (for example an adolescent who is detained for a week at juvenile detention facility) may resume research activities when he/she is no longer incarcerated or in a court mandated facility if the time remaining for study participation has not lapsed.
* No study procedures or activities will be conducted with any participant while he/she is incarcerated or in a court mandated facility.

Ages: 10 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 324 (Actual)
Dates: Start 2009-04; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Home visit assessment | Yearly
  Includes caregiver packets (including CBCL, Sleep Habits Questionnaire, and Modifiable Activity Questionnaire for Adolescents), child assessment (including Sleep Habits Questionnaire, Modifiable Activity Questionnaire for Adolescents, Children's Affective Dysregulation Scale, and Children's Affective Lability Scale) and Parent-Child videotaped discussions. Additionally, child will be fitted with a SenseWear Armband device.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Shaw, PhD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States